CLINICAL TRIAL: NCT06717503
Title: Medico-legal Aspects of Acute Spinal Injuries At Trauma Unit of Assiut University Hospital
Brief Title: Medico-legality of Acute Spinal Cord Injuries
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Khalid Mohamed Ismail, Demonstrator at forensic medicine and clinical toxicology, Assiut University
Other Study IDs: Acute spinal cord injuries
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: data collection — data will be collected from data sheets of acute spinal cord injury patients (Patients' demographic and epidemiological ,Mode of trauma, Cause of injury, Method of arrival to hospital, Time passed between trauma and arrival at hospital,How to deal with the TSI patients from the time of the injury until arrival at hospital, Examination findings, Imaging findings, Type and level of the injury, Sequels, Hospital stay period and operations)

SUMMARY:
1. Describe different medico-legal aspects of TSI (mode of trauma, cause and Pattern of spinal injuries).
2. Assess the outcome of TSI in studied cases.
3. Associate type of trauma with the different patterns of acute spinal injuries.

DETAILED DESCRIPTION:
A medico-legal case (MLC) applies to any case of injury or medical condition in which law enforcement agencies seek to investigate and fix the responsibility regarding the said injury or medical condition. From a physician's perspective, a MLC is a medical or clinical case with legal implications. In such cases presented directly to the hospital, after obtaining a detailed history and examination of the patient, the physician concludes the need for the law enforcement administration to investigate further. Besides, such cases could also be referred to the physician by the law enforcement administration for application of medical expertise and opinion to aid in the administration of justice .

Trauma is the 6th leading cause of death worldwide resulting in 5 million of all deaths. It is the 5th leading cause of significant disability . In Egypt, injuries the fifth leading cause of death and the most common cause of hospitalization and account for at least 1/4 of all inpatient(World Health Organization 2009). Spine is one of the body parts that is commonly subjected to trauma . Traumatic spinal injuries as seen from a medico-legal point of view, is an integral part of medical practice in emergency department..

SCI is associated with permanent disability and decreased life expectancy .Although more than 80% of the world's population live in the more than 100 developing countries, little information is available regarding the epidemiology of SCI in these countries . The higher prevalence of TSI may be due to the increased frequency of events causing injury, such as road traffic accidents (RTAs), and higher rates of occupational-related incidents, such as falls from trees .

Permanent infirmity is a major sequel of spinal fractures, it is considered as a legal as well as a medical problem. Physician should be oriented about the legal issues of compensation to help them in saving patients' rights . The cervical spinal cord is the most commonly affected level, followed by the thoracic and lumbar . Lower thoracic lesions can cause paraplegia while lesions at cervical level are associated with quadriplegia.

Concerning the mechanisms of injury, they differ in different age groups: common causes are road accidents, followed by traumas caused by falls, attacks, sports, or occupational-related Incidents . Imaging investigations showing different types of spinal cord injuries including fracture, dislocation, damage to the intervertebral discs, ligament tear, vascular affection, and associated injures . TSI occurs more frequently and has worse outcomes in low and middle-income countries than in high-income countries .

The number of disabled has increased considerably. The development constitutes a good reason for paying more specific attention to society's growing number of disabled. To our knowledge, up to 2024 there is a deficient studies in medico-legal aspect of traumatic spinal injuries and its squeals in Upper Egypt.

ELIGIBILITY:
Inclusion criteria:

* All patients presenting with acute TSI regardless level of injury, or neurological status.

Exclusion criteria:

* Patients have congenital anomalies, neurological defects or disability before trauma.
* Patients with pathological spinal cord diseases were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A structured data sheet is prepared and included the following:
  (A)Patients' demographic and epidemiological data such as age, sex, residence, education and marital state.
  (B)Mode of trauma (accidental, homicidal, suicidal). (C)Cause of injury like motor car, motor cycle accident, fall from height, blunt trauma, sports, occupation….etc.
  (D)Method of arrival to hospital. (E)Time passed between trauma and arrival at hospital. (F)How to deal with the TSI patients from the time of the injury until arrival at hospital.
  (G)Examination findings, including careful documentation of the neurological status.
  (H)Imaging findings, including plain X-rays, MSCT, and MRI. (I)Type and level of the injury (fracture, dislocation, ligament tear, associated bone injuries…etc).
  (J)Sequels (deformity, disability, permanent infirmity and death). (K)Hospital stay period and operations
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of medico-legal aspects of traumatic spinal injury cases includind 1 mode of trauma: suicidal, homicidal or accidental 2 causes :road traffic injuries, fall from height, assault from other...etc 3 Pattern: type and level of the injury. | baseline
  A structured data sheet is prepared and included the following:
  (A)Patients' demographic and epidemiological data such as age, sex, residence, education and marital state.
  (B)Mode of trauma (accidental, homicidal, suicidal). (C)Cause of injury like motor car, motor cycle accident, fall from height, blunt trauma, sports, occupation….etc.
  (G)Examination findings, including careful documentation of the neurological status.
  (H)Imaging findings, including plain X-rays, MSCT, and MRI. (I)Type and level of the injury (fracture, dislocation, ligament tear, associated bone injuries…etc).
  (J)Sequels (deformity, disability, permanent infirmity and death). this data will be collected from the patients and analysis to data

SECONDARY OUTCOMES:
Determine the association between causes of trauma( motor car, motor cycle accident, fall from height, blunt trauma, sports, occupation….etc) with the different patterns of acute spinal injuries including type and level from imaging investigation. | baseline
  after analysis of data we will make a correlation between the data like Determine the association between causes of trauma( motor car, motor cycle accident, fall from height, blunt trauma, sports, occupation….etc) with the different patterns of acute spinal injuries including type :fracture or dislocation and level :cervical or lumber from imaging investigation .

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Mohamed Abd El Rahman, Assistant Professor, Study Director — Doaa Mohamed Abd El Rahman; Ali Mohamedein Mohamed, professor, Study Director — Ali Mohamedein Mohamed

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson JR, Cadotte DW, Fehlings MG. Clinical predictors of neurological outcome, functional status, and survival after traumatic spinal cord injury: a systematic review. J Neurosurg Spine. 2012 Sep;17(1 Suppl):11-26. doi: 10.3171/2012.4.AOSPINE1245. PMID 22985366
- [Background] Vazquez XM, Rodriguez MS, Penaranda JM, Concheiro L, Barus JI. Determining prognosis after spinal cord injury. J Forensic Leg Med. 2008 Jan;15(1):20-3. doi: 10.1016/j.jflm.2007.06.003. Epub 2007 Sep 25. PMID 18096510
- [Background] Singh A, Tetreault L, Kalsi-Ryan S, Nouri A, Fehlings MG. Global prevalence and incidence of traumatic spinal cord injury. Clin Epidemiol. 2014 Sep 23;6:309-31. doi: 10.2147/CLEP.S68889. eCollection 2014. PMID 25278785
- [Background] Soreide K. Epidemiology of major trauma. Br J Surg. 2009 Jul;96(7):697-8. doi: 10.1002/bjs.6643. No abstract available. PMID 19526611
- [Background] Kumar R, Lim J, Mekary RA, Rattani A, Dewan MC, Sharif SY, Osorio-Fonseca E, Park KB. Traumatic Spinal Injury: Global Epidemiology and Worldwide Volume. World Neurosurg. 2018 May;113:e345-e363. doi: 10.1016/j.wneu.2018.02.033. Epub 2018 Feb 14. PMID 29454115
- [Background] Blackmore CC, Emerson SS, Mann FA, Koepsell TD. Cervical spine imaging in patients with trauma: determination of fracture risk to optimize use. Radiology. 1999 Jun;211(3):759-65. doi: 10.1148/radiology.211.3.r99jn22759. PMID 10352603
- [Background] Aktas N, Gulacti U, Lok U, Aydin I, Borta T, Celik M. Characteristics of the Traumatic Forensic Cases Admitted To Emergency Department and Errors in the Forensic Report Writing. Bull Emerg Trauma. 2018 Jan;6(1):64-70. doi: 10.29252/beat-060110. PMID 29379812